CLINICAL TRIAL: NCT04862962
Title: Retrospective Study to Evaluate the Safety of the Fixed-dose Combination Rosuvastatin / Ezetimibe as a Treatment for Patients With Dyslipidaemia in Usual Medical Practice.
Brief Title: Study to Evaluate the Safety of the Fixed-dose Combination Rosuvastatin/Ezetimibe for Patients With Dyslipidaemia
Acronym: TREZETE
Status: Completed | Type: Observational
Sponsor: Laboratorios Silanes S.A. de C.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: SIL-30231-IV-20(1)
Record Dates: First submitted 2021-04-23; First posted 2021-04-28 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Dyslipidemias
Keywords: Dyslipidemias; Combine therapy; Lower Cholesterol; Lipids
MeSH Terms: conditions — Dyslipidemias | interventions — Ezetimibe

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group A: Rosuvastatin /Ezetimibe fixed dose (TREZETE®): Rosuvastatin /Ezetimibe fixed dose (TREZETE®) Pharmaceutical Form: Tablets Dosage: 10 mg / 10 mg or 20 mg / 10 mg Administration way: Oral
  Interventions: Drug: Rosuvastatin 10 or 20mg /Ezetimibe 10 mg Fixed Dose

INTERVENTIONS:
Drug: Rosuvastatin 10 or 20mg /Ezetimibe 10 mg Fixed Dose — Oral Tablets 10 mg/10 mg or 20 mg/10 mg
  Other Names: (TREZETE®)

SUMMARY:
Retrospective, analytical, longitudinal, multicenter study to evaluate the safety of the fixed-dose combination of rosuvastatin / ezetimibe as treatment for patients with dyslipidemia in routine medical practice.

DETAILED DESCRIPTION:
To assess the safety of the fixed-dose combination of rosuvastatin / ezetimibe in subjects older than 18 years of age (gender indistinct) with dyslipidemia who at the discretion have been candidates for treatment with the combination. For the safety analysis, all the research subjects who have taken rosuvastatin / ezetimibe will be considered. The information recorded by the treating physicians in the file will be reviewed and within the case report format (CRF) of all adverse events that occur in the study. The terms originally used in the case report format by the investigators to identify adverse events (AE) will be coded in the analysis stage of Results using the current MEdDRA dictionary. The incidence of AE will be synthesized such as the frequency count and percentage of research subjects with events adverse by organ / system.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years of age.
* Diagnosis of dyslipidemia.
* That treatment with the fixed-dose combination of rosuvastatin / ezetimibe is documented.
* Have security questioning on at least two occasions.

Exclusion Criteria:

* Subjects who has taken any other statins, fibrates, bile acid sequestrants, niacin (> 500 mg) or inhibitors of PCSK9 concomitantly during treatment with rosuvastatin / ezetimibe.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects over 18 years of age (gender indistinct) with dyslipidemia who, at the discretion of thetreating physician have been candidates for treatment with the fixed-dose combination of rosuvastatin-ezetimibe.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Adverse events presented | 2 months
  Describe the frequency and intensity of adverse events presented.
Average difference in lipid profile values | Baseline, 2 months
  Evaluate the average difference in lipid profile values between at least 2 measurements.

SECONDARY OUTCOMES:
Adherence to treatment | 2 months
  To assess adherence to treatment with rosuvastatin / ezetimibe fixed-dose combination by pill count.
Significant reduction in LDL cholesterol | 2 months
  To assess the proportion of subjects who achieved a significant reduction in LDL cholesterol at each concentration of treatment.
Percentage of patients who met established goals according to cardiovascular risk | 2 months
  To identify the percentage of patients who met the established goals according to cardiovascular risk determined by the European Society of Cardiology (ESC) and / or American Heart Association (AHA) / American College of Cardiology (ACC) recommendations.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Rodriguez Saldaña, M.D, Principal Investigator — Resultados Médicos, desarrollo e Investigación; Francisco G Padilla Padilla, M.D, Principal Investigator — Independent; Ernesto G Cardona Muñoz, M.D, Principal Investigator — Independent; David Cardona Müller, M.D, Principal Investigator — Independent; Marcos Ibarra Flores, M.D, Principal Investigator — Cardiólogos Certificados S.C; José A Estrada Suarez, M.D, Principal Investigator — Independent
Locations (1):
- Laboratorio Silanes, S.A. de C.V., Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garcia-Garcia G, Aviles-Gomez R, Luquin-Arellano VH, Padilla-Ochoa R, Lepe-Murillo L, Ibarra-Hernandez M, Briseno-Renteria G. Cardiovascular risk factors in the Mexican population. Ren Fail. 2006;28(8):677-87. doi: 10.1080/08860220600936096. PMID 17162426
- [Background] Roth GA, Fihn SD, Mokdad AH, Aekplakorn W, Hasegawa T, Lim SS. High total serum cholesterol, medication coverage and therapeutic control: an analysis of national health examination survey data from eight countries. Bull World Health Organ. 2011 Feb 1;89(2):92-101. doi: 10.2471/BLT.10.079947. Epub 2010 Sep 3. PMID 21346920
- [Background] Escobedo-de la Pena J, de Jesus-Perez R, Schargrodsky H, Champagne B. [Prevalence of dyslipidemias in Mexico city and Its relation to other cardiovascular risk factors. Results from the CARMELA study]. Gac Med Mex. 2014 Mar-Apr;150(2):128-36. Spanish. PMID 24603993
- [Background] Adhyaru BB, Jacobson TA. Safety and efficacy of statin therapy. Nat Rev Cardiol. 2018 Dec;15(12):757-769. doi: 10.1038/s41569-018-0098-5. PMID 30375494
- [Background] Luvai A, Mbagaya W, Hall AS, Barth JH. Rosuvastatin: a review of the pharmacology and clinical effectiveness in cardiovascular disease. Clin Med Insights Cardiol. 2012;6:17-33. doi: 10.4137/CMC.S4324. Epub 2012 Feb 1. PMID 22442638
- [Background] Cheng JW. Rosuvastatin in the management of hyperlipidemia. Clin Ther. 2004 Sep;26(9):1368-87. doi: 10.1016/j.clinthera.2004.09.005. PMID 15531000
- [Background] Rubba P, Marotta G, Gentile M. Efficacy and safety of rosuvastatin in the management of dyslipidemia. Vasc Health Risk Manag. 2009;5(1):343-52. doi: 10.2147/vhrm.s3662. Epub 2009 Apr 8. PMID 19436657
- [Background] Kones R. Rosuvastatin, inflammation, C-reactive protein, JUPITER, and primary prevention of cardiovascular disease--a perspective. Drug Des Devel Ther. 2010 Dec 9;4:383-413. doi: 10.2147/DDDT.S10812. PMID 21267417
- [Background] Battaggia A, Donzelli A, Font M, Molteni D, Galvano A. Clinical efficacy and safety of Ezetimibe on major cardiovascular endpoints: systematic review and meta-analysis of randomized controlled trials. PLoS One. 2015 Apr 27;10(4):e0124587. doi: 10.1371/journal.pone.0124587. eCollection 2015. PMID 25915909
- [Background] Ballantyne CM, Weiss R, Moccetti T, Vogt A, Eber B, Sosef F, Duffield E; EXPLORER Study Investigators. Efficacy and safety of rosuvastatin 40 mg alone or in combination with ezetimibe in patients at high risk of cardiovascular disease (results from the EXPLORER study). Am J Cardiol. 2007 Mar 1;99(5):673-80. doi: 10.1016/j.amjcard.2006.10.022. Epub 2007 Jan 4. PMID 17317370
- [Derived] Rodriguez-Saldana J, Padilla-Padilla F, Cardona-Munoz EG, Romero-Antonio Y, Arguedas-Nunez MM, Sander-Padilla JG, Martinez-Munoz A, Lugo-Sanchez LA, Rodriguez-Vazquez IC, Gonzalez-Canudas J. Real-World Evidence Evaluation on the Lipid Profile, Therapeutic Goals, and Safety of the Fixed-Dose Combination of Rosuvastatin/Ezetimibe (Trezete(R)) in Dyslipidemia Patients. Cardiol Res Pract. 2022 Sep 10;2022:9464733. doi: 10.1155/2022/9464733. eCollection 2022. PMID 36124294